CLINICAL TRIAL: NCT06354205
Title: Comparison of Salivary Procalcitonin (PCT) Levels and Serum PCT Levels in Infants Under 1 Year of Age Suspected of Systemic Bacterial Infection
Brief Title: Comparison of Salivary Procalcitonin (PCT) Levels and Serum PCT Levels
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Caner Turan, Caner Turan, Ege University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 24-3.1T/98
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Bacterial Infections; Children, Only; Procalcitonin; Saliva
Keywords: procalcitonin; saliva; children; infection
MeSH Terms: conditions — Bacterial Infections; Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients selection (Other): Children under 1 year of age will be recruited for saliva and blood sample collection in the study
  Interventions: Diagnostic Test: Sliva Procalcitonin

INTERVENTIONS:
Diagnostic Test: Sliva Procalcitonin — Sliva Procalcitonin vs Blood procalcitonin

SUMMARY:
Recently, it has been seen that investigations from saliva samples could be an alternative to those from blood samples. Saliva collection is a simple, non-invasive, cost-effective, and relatively easy method, making it potentially suitable as a new diagnostic tool in pediatric patients. In the current literature, elevated levels of saliva CRP, TNF-α, IL-6, and IFN-γ have been reported in inflammatory conditions. However, while there are animal studies suggesting the use of saliva PCT levels for focal diseases such as gingival inflammation and periodontitis and as a potential tool for non-invasive detection of sepsis, there is no human study regarding its use in systemic infections.

The aim of this study is to evaluate the correlation between serum PCT levels and saliva PCT levels in children suspected of SBE and to determine the diagnostic value of saliva PCT.

ELIGIBILITY:
Inclusion Criteria:

* Being under one year of age
* Having serum Procalcitonin (PCT) requested due to suspicion of systemic infection

Exclusion Criteria:

* Being over one year of age
* Having a chronic illness that could cause elevation in inflammatory biomarkers
* Taking any medication (such as antibiotics, immunomodulatory, or immunosuppressive drugs, etc.) that could affect inflammatory biomarkers
* Diagnosis of gingivostomatitis

Ages: 0 Years to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Correlation | One year
  the correlation between serum Procalcitonin (PCT) levels and salivary PCT levels

SECONDARY OUTCOMES:
Diagnose | One year
  Diagnostic value of saliva PCT

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University School of Medicine, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No